CLINICAL TRIAL: NCT05656833
Title: Combination Topical Cysteamine and Fractional 1927nm Low-Powered Diode Laser
Brief Title: Combination Topical Cysteamine and Fractional 1927nm Low-Powered Diode Laser for Treatment of Facial Melasma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UnionDerm (Other)
Collaborators: Solta Medical (Industry); Skin of Color Society (Unknown); Scientis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SterlingIRB Study #9727
Record Dates: First submitted 2022-12-06; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Melasma
Keywords: Facial Melasma; Cyspera; Clear & Brilliant Laser; Laser; Melasma
MeSH Terms: conditions — Melanosis; Margins of Excision | interventions — Cysteamine

STUDY DESIGN:
Intervention Model Description: Single Center, Prospective, With Before-After Analysis
Who Masked: Outcomes Assessor
Masking Description: Photographic assessment by two blinded dermatologists will measure changes will assess improvement in melasma by mMASI score. In addition, an investigator quartile improvement score from baseline to week 12 (0 - 0%, no improvement; 76%-100% - very significant improvement) will be assessed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fractional 1927nm Low-Powered Diode Laser combined with Topical Cysteamine (Active Comparator): One side of the face of participants will be randomized to receive fractional 1927nm Low-Powered Diode Laser in combination with topical cysteamine. There are 3 total treatments with the laser, in combination with using the topical cysteamine cream every day for the duration of the study (12 weeks)
  Interventions: Device: Fractional 1927nm Low-Powered Diode Laser; Other: Topical Cysteamine
- Topical Cysteamine Alone (Active Comparator): The other side of the face that is not randomized to receive laser treatment will be subject to treatment with the topical cysteamine cream alone. Participants will use the topical cysteamine cream every day for the duration of the study (12 weeks).
  Interventions: Other: Topical Cysteamine

INTERVENTIONS:
Device: Fractional 1927nm Low-Powered Diode Laser — Clear & Brilliant Permea® Laser used on the side of the face randomized to receive laser
  Arms: Fractional 1927nm Low-Powered Diode Laser combined with Topical Cysteamine
Other: Topical Cysteamine — Topical Cysteamine cream will be used on the entire face.

SUMMARY:
The primary objective of our study is to determine the efficacy of combined topical cysteamine cream with a 1927 diode non-ablative laser (Clear + Brilliant Permea®; Solta Medical, Inc.), compared to topical cysteamine (Cyspera) alone in the treatment of melasma.

The main questions it aims to answer are

* If melasma treatment with topical cysteamine cream is more effective when used with the Clear & Brilliant® Permea laser
* The safety & efficacy of melasma treatment in various skin types using the Clear & Brilliantt® Permea laser in combination with topical cysteamine.

Participants will

* Come into our office for an initial screening appointment to determine if participant is eligible for the study
* Come in for 3 laser treatments, 4 weeks apart, on 1 side of the face
* Use the study provided Cyspera topical cream every day on the entire face for the 12 weeks on the study.

Researchers will compare the side of the participants face not treated with laser to the side of the face treated with laser. The participants will be using Cyspera on both sides of their face.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of Skin Type I-VI females.
* Subjects must be between 18 and 74 years of age, and must have visible melasma on the face.
* Subjects must read, understand, and sign the Informed Consent.
* Subjects must be willing and able to comply with all follow-up requirements.

Exclusion Criteria:

* Subjects must not have active or localized or systemic infections.
* Subjects must not be immunocompromised.
* Subjects must not have a coagulation disorder, and must not be using anticoagulation -medications.
* Subjects must not have history of surgical or cosmetic treatment, including prior skin lightening agents, microneedling or microdermabrasion, or laser or light-based therapies, to the planned treatment areas in the prior 8 weeks.
* Subjects must not have photosensitivity or allergy.
* Subjects must not be mentally incompetent.
* Subjects must not be pregnant or breastfeeding.
* History of skin cancer or pre-cancerous lesions in the treatment area
* Subjects must not be currently using aspirin or antioxidants.
* Subjects must not refuse to sign the Informed Consent document and/or refuse to comply with all follow-up requirements.
* Subjects must never have had gold therapy.
* Subjects must never have had radiation therapy to the face. Recent or current suntan or sunburn within 2 weeks.
* Clinically dysplastic nevi in the treatment area.
* Subjects must not have had collagen, other methods of tissue augmentation, botox, chemical peels, dermabrasion, or resurfacing within the last year.
* Oral retinoid (Accutane or Soriatane) or photosensitizing drugs, e.g. Declomycin®, a tetracycline with light absorption in the range of 400 to 450 nm use within 24 months of study entry.
* Topical retinoid therapy on face within one month of study entry.
* History of keloids or hypertrophic scars
* A history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins, or photodermatosis.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The primary objective of our study is to determine the efficacy of combined topical cysteamine cream with a 1927 diode non-ablative laser (Clear + Brilliant Permea®; Solta Medical, Inc.), compared to topical cysteamine alone in the treatment of melasma. | 12 Weeks
  Photographic assessment by two blinded dermatologists will measure changes will assess improvement in melasma by modified Melasma Area and Involvement Index (mMASI). Total mMASI score ranges from 0 - 24, with a higher score indicating more involvement and/or severity of melasma

CONTACTS AND LOCATIONS:
Locations (1):
- UnionDerm, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Investigator has not decided on IPD sharing plan yet

REFERENCES:
- See also: Contact / Official Website for UnionDerm — https://www.unionderm.com/innovations/current-studies-and-clinical-trials/

DOCUMENTS (2):
  • Study Protocol (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT05656833/Prot_000.pdf
  • Informed Consent Form (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT05656833/ICF_001.pdf